



## Comitato Etico per la Ricerca

#### PROJECT TITLE

Effects of an adapted multicomponent training program (Adapted Physical and Sports Activity - AFA) for promoting mental and physical well-being in cancer survivors currently in physiological or chronic-stabilized condition.

#### LABORATORY/DEPARTMENT

Laboratory of Exercise Science and Sport, Degree Program in Sports Science and Techniques, Department of Translational Biomedicine and Neurosciences (DiBraiN), University of Bari – Aldo Moro

EXPERIMENTAL DESIGN

Interventional

EXPECTED START AND END DATE OF THE PROJECT

January 2025 – June 2025

FUNDS USED FOR THE PROJECT

No

DATE OF THE DOCUMENT

20/02/2025





Comitato Etico per la Ricerca

## INFORMED CONSENT FORM FOR PARTICIPATION IN THE STUDY/RESEARCH PROJECT

Dear Sir/Madam,

You are invited to participate in the research study/project titled "Effects of an adapted multicomponent training program (Adapted Physical and Sports Activity - AFA) for promoting mental and physical well-being in cancer survivors currently in physiological or chronic-stabilized condition". In order to make an informed decision, we are providing you with information about the nature of the study, the objectives of the project, and the activities in which you may be involved for the accomplishment of the research goals.

Please read these details carefully before deciding whether to participate in the project. You may ask any questions for clarification and raise any concerns that have not been answered clearly and thoroughly.

If, after reading and understanding all the provided information, you decide to participate in the study, you will be asked to sign and date the attached Informed Consent Form.

Your personal data will be processed as described in the specific privacy notice, in accordance with EU Regulation 2016/679 and Legislative Decree No. 196/2003. This privacy notice and the related request for consent to data processing will be provided to you separately.

**Research title**: Effects of an adapted multicomponent training program (Adapted Physical and Sports Activity - AFA) for promoting mental and physical well-being in cancer survivors currently in physiological or chronic-stabilized condition.

CUP Project: N/D Sponsor: N/D

implementing organizations: N/D

#### INFORMATION REGARDING PARTICIPATION IN RESEARCH

#### **OBJECTIVES:**

The research project aims to evaluate the effectiveness of a multicomponent training protocol (MCT) on the following parameters: psychological, physical fitness, mental well-being, and quality of life, in cancer survivors currently in a stabilized condition, compared to an aerobic training protocol (AT) and a waiting control group (WLCG). In addition, the aim is to evaluate the impact of training in participants' coping strategies, i.e., the ways in which they manage stress, emotional difficulties and daily challenges, in order to foster better psychological adaptation and greater autonomy. To achieve this objective, the researchers involved in the project aim to collect and analyze data on the estimation of these parameters through physical and psychological tests to be performed before and after the intervention.





#### Comitato Etico per la Ricerca

#### STUDY/PROJECT ARTICULATION (PHASES AND TIMELINES):

#### RECRUITMENT PHASE AND COLLECTION OF INFORMED CONSENT (1-3 months)

Presentation to participants: The informed consent will be distributed during the recruitment procedures. The consent will be collected prior to the initial assessments (T0).

#### RANDOMIZATION PHASE, INITIAL ASSESSMENTS, AND DATA COLLECTION (1-2 weeks)

After recruitment, participants will be randomly assigned to one of the three groups (MCT, AT, WLCG). Subsequently, initial assessments will be conducted, consisting of motor tests and psychological questionnaires.

#### INTERVENTION PHASE (6 months)

During this phase, participants previously randomly assigned to one of the three groups (MCT, AT, WLCG), under the supervision of field experts, will begin their activities, specifically:

- MCT group: Participants will follow an adapted multicomponent training program, which includes aerobic, resistance, and mobility/flexibility exercises;
- AT group: Participants will follow an adapted multicomponent training program, which includes aerobic exercises;
- WLCG group: Participants will not perform any structured physical activity but will continue with their usual lifestyle. They will be placed on a waiting list, guaranteeing them future participation in adapted physical activity after the intervention period.

#### FINAL ASSESSMENT PHASE AND DATA COLLECTION (1-2 weeks)

Within one week after the end of the intervention period, final assessments will be initiated, consisting of motor tests and psychological questionnaires.

**Discussion and Consent Signature:** The research team will clarify any doubts of the participants. Participants will sign the consent form after understanding the details and potential risks. A minimum of 10-30 minutes must be provided per participant.

Estimated Time: 10-30 minutes per participant.

**BENEFITS:** Participants will have access to adapted physical activity tailored to their needs, with the aim of improving psychophysical conditions related to mobility, autonomy, and self-efficacy, ultimately enhancing their quality of life, all under the supervision of field experts.

**RISKS:** Participation does not involve any risk or discomfort, except for the rare possibility of traumatic events that may occur during the course of the study.





## Comitato Etico per la Ricerca

| I, the undersigned | | born in | on, |
|---|---|---|---|
| residing at | stre | et | on, hereby |
| | D | DECLARE | |
| 4.11 | | | |
| that I have read and understoo | od the informati | on and wish to partic | espate in the proposed study. |
| | □ I confirm | □ I do not con | firm |
| | SIGNATURE | | |
| specifying that by signing it, y CONSE | | CIPATE IN THE F | |
| I declare that: ☐ I have voluntarily decided t | o participate in | the research;; | |
| ☐ I have received all the information related to the request to participate in the research, particularly regarding the purpose, procedures, and what is required of me; | | | |
| ☐ I have received, read, and understood the document containing the "Information regarding participation in the research," which was provided to me, and I have received all the necessary information for my responsible participation in the research; | | | |
| ☐ I have had the opportunity answers; | to ask question | as and have received | clear, complete, and satisfactory |
| ☐ I have been informed about | potential risks; | | |
| ☐ I am aware that my particip | ation is voluntar | y; | |
| ☐ I have been assured that I consequences on the | | | ny time, and that this will have no |

For any doubts or questions, you can contact the Dr. Alessandro Petrelli





## Comitato Etico per la Ricerca

Phone 3272744090

| Full name of the participant Signature of the participant | Date |
|-----------------------------------------------------------|----------|
| Full name of the person who obtained the consent | |
| Signature of the research supervisor | Date |
| Full name of any witnesses present | |
| Signature of the witnesses present | <br>Date |





## Comitato Etico per la Ricerca

#### WITHDRAWAL OF CONSENT

If you wish to withdraw your consent to participate in this research, please indicate with an "X" the desired option among the following:

I withdraw my consent to continue participating in one or more of the following activities (please specify the individual activities for which you wish to exercise the right to withdraw consent):

| • | |
|--------------------------------------------------|----------|
| • = | |
| • | |
| Full name of the participant | · |
| Signature of the participant | Date |
| Full name of the person who obtained the consent | <br>Date |
| rightene of the research supervisor | Bute |
| Full name of any witnesses present | |
| Signature of the witnesses present | <br>Date |





## Comitato Etico per la Ricerca

In case of incapacitated individuals and minors:

# CONSENT DECLARATION FOR THE PROCESSING OF PERSONAL DATA OF THE SUBJECT CONCERNED BY THE PARENT/GUARDIAN/ CURATOR/ SUPPORT ADMINISTRATOR

# PURSUANT TO AND FOR THE PURPOSES OF THE EUROPEAN DATA PROTECTION REGULATION

| I, the | undersigned | , born on |
|---|---|---|
| | in | |
| in the cap | acity of □ guardian □ curator □ support administrator of | |
| (name) _ | (surname)in | , born on |
| in accorda | ance with the provisions of Regulation (EU) 2016/679 and Legislative Decreat amendments and integrations, and having read the "Information on the | ee 196/2003 and |
| | ☐ I consent ☐ I do not consent | |
| person con | cessing - necessary for participation in the research in question - of the personcerned, including health-related data, for scientific and statistical research and for the reasons described in the section titled "Purpose and methods of described in the section titled". | purposes, in the |
| | ☐ I consent ☐ I do no consent | |
| | rage and further use — not necessary for participation in the study in question e person concerned for subsequent research activities and to be possibly cont | _ |
| Additiona | ally, I consent I do not consent | |
| other aud | occessing of images of the person concerned (video, audio, and photograph iovisual materials) - necessary for participation in the study - for the rein point (4.A) and in compliance with copyright law. | • |
| Date | Signature | |